CLINICAL TRIAL: NCT04420780
Title: Study Protocol for a Randomized Clinical Trial to Evaluate the Effect of the Use of Xylitol Gum in the Prevention of Caries Lesions in Children Living in Ladakh - the Caries Prevention Xylitol in Children (CaPreXCh) Trial
Brief Title: Effect of the Use of Xylitol Gum in the Prevention of Caries Lesions in Children Living in Ladakh
Acronym: CaPreXCh
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the political sistuation the recruitment was withdrawn
Sponsor: University of Bern (Other)
Collaborators: University of Milan (Other); Università degli Studi di Sassari (Other); WHO Collaborating Center for Epidemiology and Preventive Dentistry (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CaPreXCh
Record Dates: First submitted 2020-05-25; First posted 2020-06-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Caries
Keywords: Caries prevention; Xylitol gum; Children
MeSH Terms: interventions — Xylitol; Sweetening Agents

STUDY DESIGN:
Intervention Model Description: This is a triple-blind randomized, controlled, parallel-group clinical trial. Two groups will be compared: subjects who will receive a 100% xylitol chewing gum, and those who will receive a 22% xylitol gum.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xyl Group (Experimental): Children will receive sugar-free gums containing 100% Xylitol as sweetener
  Interventions: Dietary Supplement: Administration of sugar-free gums sugar-free gums containing 100% Xylitol as sweetener
- Pol Group (Active Comparator): Children will receive sugar-free gums containing a polyols mixture plus a low amount of Xylitol (22%).
  Interventions: Dietary Supplement: Administration of sugar-free gums sugar-free gums containing containing a polyols mixture plus a low amount of Xylitol (22%)

INTERVENTIONS:
Dietary Supplement: Administration of sugar-free gums sugar-free gums containing 100% Xylitol as sweetener — The subjects will be instructed to chew a total of 6 pellets for 5 min divided into 3 intakes a day (2 in the morning, 2 after the midday meal and 2 in the afternoon)
  Arms: Xyl Group
Dietary Supplement: Administration of sugar-free gums sugar-free gums containing containing a polyols mixture plus a low amount of Xylitol (22%) — The subjects will be instructed to chew a total of 6 pellets for 5 min divided into 3 intakes a day (2 in the morning, 2 after the midday meal and 2 in the afternoon)
  Arms: Pol Group

SUMMARY:
Background: Ladakh is a region administered by India, covering an area slightly larger than Croatia; it is part of the larger region of Kashmir and Jammu. Till now, oral health data on population living in Ladakh are not available. The aim of the present preventive project will be to record the caries prevalence of schoolchildren living in Ladakh and to implement a school-based xylitol program using chewing gums in order to reduce caries incidence.

Methods: The protocol of the Caries Prevention Xylitol in Children (CaPreXCh) trial is designed as a triple-blind randomized, controlled, parallel-group clinical trial in children aged 5-14 years. The study will be carried out from August 2021 to August 2024 in Zanskar Valley (Ladakh). Participants will be randomly allocated into two groups: subjects who will receive a 100% xylitol chewing gum, and those who will receive a 22% xylitol gum. The subjects will be instructed to chew a total of 6 pellets for 5 min divided into 3 intakes a day (2 in the morning, 2 after the midday meal and 2 in the afternoon) for one school-year. Clinical examination will comprise an oral examination: caries index (ICDAS scores), bleeding on probing recording and evaluation of plaque pH fluctuation after sucrose challenge and will be performed at baseline (t0) and repeated 12 months at the end of the chewing-gum administration period (t1) as interim examination, after 12 months (t2) and 24 months (t3) after the end of the experimental period (chewing gum use). The primary outcome will be the caries increment measured both at enamel and dentinal level. Data analysis will be conducted through Kaplan-Meyer graphs to evaluate caries increment as primary outcome, and the methods will be compared to each other with Cox regression with shared frailty. The net caries increment for initial, moderate and severe caries level, using ICDAS (Δ-initial, Δ-moderate and Δ-severe), will be calculated.

Discussion: This is the first clinical trial to assess the effect of chewing gum containing only xylitol as sweeteners for caries prevention. Moreover, the children object of this study is a population with special living conditions.

DETAILED DESCRIPTION:
The study will be carried out from August 2021 to August 2024 in Zanskar Valley (Ladakh).

Participants, interventions and outcomes Setting The study will be conducted in the Zanskar Valley (Ladakh). The subjects (5 to 14 years old) will be randomly selected from a list of school class in the selected schools.

Interventions

After obtaining actual caries data, schools with similar numbers of schoolchildren (at least 300 subjects per school) will be selected for the preventive project. The participants will be randomly taking as cluster the school-class allocated into two groups (Figure 1). Randomization will be performed by one author (G. Campus) using Microsoft Excel for Mac (version 16.37) in permuted blocks of 2 or 4 with a random variation of the blocking number, and 2 groups will be created:

1. the first group (Xyl) will receive sugar-free gums containing 100% Xylitol as sweetener;
2. the second group (Pol) will receive sugar-free gums containing a polyols mixture plus a low amount of Xylitol (22%).

   All chewing gums will be produced and supplied by Perfetti Van Melle SpA (Lainate, Italy). The xylitol chewing gum is with xylitol (64% w/v) as the only sweetener. The polyols chewing gum is a sugar-free gum with 22% of Xylitol, 30% Sorbitol, 6% Maltitol syrup and 4% Mannitol. All types of chewing gums weigh 1.4 g each and will be identical in colour, shape and taste. The treatment will follow the school year calendar for a total of nine months of administration.

   Clinical examination

   Clinical examination will comprise an oral examination (caries index, bleeding on probing recording) and evaluation of plaque pH fluctuation after sucrose challenge. Bleeding on probing will be used as a proxy of plaque presence, since there is a causal relationship between bleeding on probing and amount of plaque.

   The subjects will be examined using a mouth mirror, a ball ended probe and artificial light in a dental chair. Caries registration will be performed with regard to the first and second primary, and first and second permanent, molars. The International Caries Detection and Assessment System (ICDAS) will be use to record caries at tooth level as initial or moderate or severe lesions, the number of filled teeth and the missing teeth for caries. Initial caries lesion can be defined as a primary lesion, which has not reached the stage of an established lesion with cavitation (ICDAS score 1 and 2). Moderate caries lesions are defined as white or brown spot lesion with localized enamel breakdown or an underlying dentine shadow without visible dentine exposure (ICDAS score 3 and 4). Severe caries lesions are defined as distinct cavity in opaque or discoloured enamel with visible dentine (ICDAS score 5 and 6). The bleeding on probing score will be registered in all subjects.

   Plaque-pH measurements

   Interproximal-plaque pH will be evaluated using pH indicator strips , which measure a pH value in the range of 4.0-7.0 (Spezialindikator, pH range 4.0-7.0; Merck, Darmstadt, Germany). The strips determine changes in plaque pH, discriminating differences at the level of 0.2-0.5 pH units and they are easy to use. The strips are cut into 4 pieces (approx. 2 mm in width) in order to get a strip that could be easily inserted into the interproximal space and held in situ for 10 s, and its colour compared to the colour index scheme supplied by the manufacturer.

   For each subject, 3 measurements will be carried out in 2 sites, between the 2nd premolar or the 2nd primary molar, if present, and the 1st molar right and left of the upper jaw. Measurements will be performed before and at 2, 5, 10, 15, 20 and 30 min after a mouth rinse with 10% sucrose.

   Calibration of the examiners

   Prior the start of the examiners that performed all the dental screenings was trained and calibrated by a benchmark examiner. Baseline training consists in one-day theoretical course, followed by examination on extracted teeth plus a session of photographs of extracted teeth. After two days of the theoretical course a clinical training will be performed. The children were re-examined after 72 h. Inter-examiner reliability with the benchmark examiner will be evaluated using fixed-effects analysis of variance and intra-examiner reproducibility assessed as the percentage of agreement using Cohen's kappa statistic.

   Treatment

   The subjects will be instructed to chew a total of 6 pellets for 5 min divided into 3 intakes a day (2 in the morning, 2 after the midday meal and 2 in the afternoon). Thus, the total daily intake of xylitol in the Xyl group is fixed in 5.4 g and 1.8 g in the Pol group. Subjects will be instructed to use the chewing gum immediately after main meals and snacks. To the parents/guardians will be not requested to make changes in dietary and oral hygiene habits of their children. Tooth brushing will be not allowed for at least 1 h after the chewing gum use. All subjects will receive a fluoridated toothpaste containing 1,450 mg/g NaF and a manual toothbrush to be used during the experimental period, that will be supplied during the entire experimental period (2 years). All children will be instructed to brush teeth twice a day (after breakfast and supper) for 2 minutes using vertical movements.

   In order to evaluate the success of the administration of chewing gum at school, teachers will receive chewing gums necessary for a single month at a time. Children will have to return the empty blister packs when receiving those for the following month. This procedure will be repeated for all experimental (chewing) period (1-year school calendar/9 months).

   Outcomes

   The primary outcome will be the caries increment measured both at enamel and dentinal level. The secondary outcomes will be the differences obtained comparing caries increment and the variation of plaque pH in relation to the treatment decision. Furthermore, a cost- effectiveness analysis will be performed using as outcome measure the quality-adjusted life years (QALY).

   Participant timeline

   The study will be recruiting patients from August 2021 to September 2022. Each subject will be enrolled for 36 months, estimating 9 months (one school year) of treatment and 27 months of follow-up.

   Recruitment

   The recruitment will occur in Zanskar Valley (Ladakh): in Padum city.

   Assignment of interventions

   Allocation: sequence generation and concealment mechanism The random list will be generated using a computer program (Microsoft Excel for Mac); the randomization will be carried out on a school-class based by G.C. in permuted blocks of 2 or 4 with a random variation of the blocking number, and 2 groups will be created.

   Chewing gums will be supplied in plain white containers coded as 'green' or 'blue' according to the group. The code is sealed by an independent monitor and not broken until the statistical analysis will be finalized.

   Implementation

   All examinations of the children enrolled will be done by calibrated examiners. The clinical examination of the enrolled sample will be performed at baseline (t0) and repeated 12 months at the end of the chewing-gum administration period (t1) as interim examination, after 12 months (t2) and 24 months (t3) after the end of the experimental period (chewing gum use).

   Blinding

   All personnel involved into the study will be blinded to the participant assignment.

   Children, parents/caregivers and teachers responsible for the treatment, examiners who will evaluate the outcomes and statistician who will analyse data will be blind to the allocation group of the participants.

   Data collection, management, and analysis

   The follow-up assessments will be performed by a pre-calibrated blind examiner. The clinical data will be recorded on electronic sheets organized on PageMaker and then transferred to Microsoft Excel Software. The data will be cleaned, deleting those revealing the participants' identities, will be share in a public repository at the moment of the submission of the manuscripts.

   Data on caries will be based considering the tooth as the unit of analysis; the net caries increment for initial, moderate and severe caries level, using ICDAS (Δ-initial, Δ-moderate and Δ-severe), will be calculated in primary and permanent molars. Differences between groups in terms of the caries increment will be evaluated using the nonparametric Mann-Whitney U test. Kaplan-Meyer graphs will be constructed to evaluate caries increment as primary outcome, and the methods will be compared to each other with Cox regression with shared frailty. The calculation of sensitivity, specificity and accuracy will consider the results obtained with the indices and the classification of the presence or not of caries lesion by the proposed reference standard. The cost-effectiveness ratio will also be verified, considering as effect, the prevention of the primary outcome. For all tests, two-tailed analyses will be used, considering a level of significance of 5%. The quality-adjusted life-year index (QALY) will be calculated to assess the value of the preventive interventions.To determine QALYs, the utility value associated with a given state of health by the years lived in that state will be calculated. A year of life lived with no caries increment will be worth 1 QALY (1 year of life × 1 Utility value].

   Analyses will be performed using the statistical package Stata 16.0 (Stata Corp, College Station, USA).

   Monitoring

   Data monitoring An independent regulation of data collection, management and analysis will be assumed independently by the authors.

   Harms

   The procedures performed offer minimal risk to oral health of patients. Side effects of the administration of both chewing gums will be assessed by means of a questionnaire administered to the participants' parents after 3 months from the beginning of the experimental period and a second time at the end of the administration (1 year after the baseline).

   Auditing

   The data entered will be conducted by one of the authors of the study. The data will be weekly inspected. The inconsistencies will be verified, corrected and registered.

   Ethics and dissemination

   Research ethics approval, Consent and Assent

   No official Ethical committee is present in the area of the survey. The study proposal was submitted to the authorities of the Zanskar Tibetan Hospital Health Care & Sowa Rigpa Research Institute and its coordinator the Lama Zopta gave the approval for the study. Each school involved in the survey gave also the approval. Due to language problems and the low literacy rate of the population, verbal approval will be obtained for children's participation by parents or guardians.

   Confidentiality

   Participants will be coded with identification numbers to guarantee confidentiality during data analysis. Participants files will be stored in a secure room in the Department of Restorative, Preventive and Pediatric Dentistry, University of Bern.

   Access to data

   Clinical trial data will be granted full access via public repository after acceptance of the manuscripts.

   Ancillary and post-trial care

   Parents/caregivers of the children participating the trial will receive information about the children oral health.

   Dissemination policy

   A full report of the findings will be prepared and submit in full through national and international journals, newsletters and via website.

ELIGIBILITY:
Inclusion Criteria:

1. Are aged from 5 to 14 years;
2. To be in good general health;
3. Written informed consent (by the child / parent)

Exclusion Criteria:

1. Children who refuse to participate in the research; parents/guardians who refuse the participation of their children to the trial;
2. Children who present systemic conditions or chronic diseases that require differentiated care and follow-up.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline caries status in enamel (ICDAS index) | 3 years
  The primary outcome will be the caries increment measured both at surface and tooth level using ICDAS index
Change from Baseline caries status in dentine (ICDAS index) | 3 years
  The primary outcome will be the caries increment measured both at surface and tooth level using ICDAS index

SECONDARY OUTCOMES:
Plaque pH measurements in relation to the treatment decision. (PlaquepH strips) | 3 years
  Variation of plaque pH samples after sucrose challenge in relation to the treatment decision.

OTHER OUTCOMES:
Cost- effectiveness analysis | After 36 months
  Cost- effectiveness analysis using as outcome measure the quality-adjusted life years (QALY)

CONTACTS AND LOCATIONS:
Overall Officials: Guglielmo Campus, Principal Investigator — University of Bern
Locations (1):
- Moscou University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The study protocol Summer 2020/2024 Statistical Analysis Plan 2022 Analytic Code at the end of the study 2024

REFERENCES:
- [Derived] Cagetti MG, Cocco F, Calzavara E, Augello D, Zangpoo P, Campus G. Study protocol for a randomized clinical trial to evaluate the effect of the use of Xylitol gum in the prevention of caries lesions in children living in Ladakh-the Caries Prevention Xylitol in Children (CaPreXCh) trial. Trials. 2021 Dec 4;22(1):871. doi: 10.1186/s13063-021-05828-y. PMID 34863260